CLINICAL TRIAL: NCT02860091
Title: Blood Ropivacaine Concentrations Following Unilateral Chest Wall Nerve Block and Continuous Infusion in Infants and Toddlers Undergoing Thoracotomies
Brief Title: Blood Ropivacaine Concentrations Following Chest Wall Nerve Block Continuous Infusion
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Roland Brusseau, Instructor, Boston Children's Hospital
Other Study IDs: IRB-P00022295
Record Dates: First submitted 2016-08-03; First posted 2016-08-09 (Estimated); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Pain, Postoperative
Keywords: ropivacaine infusion; regional anesthesia; paravertebral block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Post-analysis specimens will be frozen and retained for further analysis, if necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ropivacaine infusion: Patients receiving continuous ropivacaine infusion for approximately 7 days via paravertebral nerve block or erector spinae catheter managed according to existing institutional protocols.
  Interventions: Drug: Ropivacaine infusion

INTERVENTIONS:
Drug: Ropivacaine infusion — Delivered via paravertebral nerve block catheter.
  Other Names: Naropin

SUMMARY:
The main objective of this proposed investigation is to evaluate blood ropivacaine concentrations in infants and toddlers following the initiation of, and over the course of, continuous paravertebral nerve blockade using ropivacaine infusion for postoperative pain control following esophageal atresia repair procedures that include posterior tracheopexy.

Continuous unilateral chest wall nerve blockade (CUCWNB) using ropivacaine is the current standard of practice for this surgical population at the investigators' institution and, as such, this study does not aim to alter the current standard clinical care received by participants but rather evaluate the blood concentrations of ropivacaine as it is routinely used.

DETAILED DESCRIPTION:
Post-surgical pain management is often suboptimal in pediatric patients, especially in those with complex past medical and past surgical histories. Physicians generally, and physicians at Boston Children's Hospital (BCH), in particular, are employing regional anesthetic techniques as either primary or adjunct measures for perioperative pain control. One of the benefits of regional anesthesia is the avoidance, or at least limitation of, opioid and benzodiazepine exposure.

CUCWNB is a regional anesthesia technique that uses an indwelling catheter, placed under ultrasound guidance, which terminates in the paravertebral space for a paravertebral nerve block or at the base of the erector spinae muscle complex immediately lateral to the paravertebral space for an erector spinae nerve block. Introduction of local anesthetic through this catheter produces ipsilateral somatic and sympathetic nerve blockade in multiple contiguous dermatomes. The technique provides effective analgesia for unilateral thoracic and abdominal surgical procedures.

CUCWNB using ropivacaine is used regularly at this institution for patients of all ages as a part of various multimodal intra- and post-operative pain management strategies. The success of CUCWNB implementation for infants and toddlers undergoing thoracotomies has been so marked that this technique has become essentially a de facto standard of care for this population at BCH.

Unfortunately, even as of today, studies demonstrating the pharmacokinetic profile of ropivacaine CUCWNB in infants and toddlers are not available. A few studies have examined plasma levels of ropivacaine after single injection paravertebral nerve blocks in adult patients. For example, a single bolus injection of 2mg/kg was well tolerated, not exceeding peak plasma concentrations of 2.5 µg/ml, well below the concentration considered a threshold for ropivacaine local anesthetic systemic toxicity (LAST). However, it is unclear how applicable this data is to our complex pediatric surgical patients at BCH.

In order to more fully understand plasma ropivacaine concentrations during CUCWNB, and particularly how these concentrations relate to known thresholds for ropivacaine-induced systemic local anesthetic toxicity, the investigators plan to measure plasma concentrations of ropivacaine at various time points following initiation of CUCWNB in infant and toddler patients having just undergone esophageal atresia repair with posterior tracheopexy.

This study does not aim to alter the current standard clinical care received by participants. No additional treatments will be provided as part of the study. Continuous ropivacaine infusion via paravertebral nerve block catheter, the standard practice for this surgical population at the investigators' institution, will be administered to enrolled (and non-enrolled) patients undergoing esophageal atresia repair with posterior tracheopexy. Paravertebral ropivacaine infusion is directed by BCH Pain Treatment Service, using existing dosage and management protocols.

The investigators' goal is to better understand plasma ropivacaine levels during continuous infusion and how they relate to currently understood thresholds for induced systemic local anesthetic toxicity in infants and toddlers, so as to develop evidence-based safety guidelines for ropivacaine infusion in infants and toddlers undergoing CUCWNB.

The investigators expect to describe the pharmacokinetics of ropivacaine via CUCWNB for postoperative pain management of infants and toddlers following thoracotomies. Knowledge of the systemic absorption of ropivacaine delivered by CUCWNB may provide new insights into appropriate dosing in order to prevent LAST. This is of particular interest in the subgroup of infants for whom rates of metabolism and elimination of local anesthetic drugs are poorly understood.

ELIGIBILITY:
Inclusion Criteria:

* Infants and toddlers (0-4) years
* Undergoing a procedure that requires a thoracotomy for esophageal atresia repair and related procedures
* Receiving ropivacaine via continuous paravertebral nerve block catheter or erector spinae catheter

Exclusion Criteria:

* Hepatic dysfunction
* Local anesthetic allergy

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients undergoing surgical esophageal atresia repair and/or related procedures receiving continuous ropivacaine via paravertebral catheter or erector spine catheter.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Blood ropivacaine concentration | 7 days
  Plasma ropivacaine concentration

CONTACTS AND LOCATIONS:
Overall Officials: ROLAND BRUSSEAU, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children"S Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No